CLINICAL TRIAL: NCT06627010
Title: Herpes Simplex Meningo Encephalitis Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, HESS Valentin, CCAH Dr, Central Hospital, Nancy, France
Other Study IDs: 2023PI237
Record Dates: First submitted 2024-01-26; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-01

CONDITIONS: Herpes Simplex Meningo Encephalitis
MeSH Terms: conditions — Encephalitis, Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: description — study of file

SUMMARY:
study of risk factors and prognosis of herpes simplex encephalitis recurrence.

ELIGIBILITY:
Inclusion Criteria:

* documented herpes simplex recurrence

Exclusion Criteria:

* other cause

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Herpes Simplex Meningo Encephalitis Recurrence
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
survival rate | 1 year
  prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Valentin HESS, Principal Investigator — CHRU NANCY
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No
anonymous